CLINICAL TRIAL: NCT05239676
Title: Clinical Study on the Safety and Effectiveness of Autologous Hematopoietic Stem Cell Transplantation Combined With CAR-T Cells in the Treatment of Refractory and Relapsed Malignant Lymphoma
Brief Title: Autologous Hematopoietic Stem Cell Transplantation Combined With CAR-T Cells in the Treatment of Refractory and Relapsed Malignant Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO-CART-001
Record Dates: First submitted 2021-12-01; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma
Keywords: ASCT; CD19 CAR-T
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of Lymphoma (Experimental): Refractory and relapsed malignant lymphoma
  Interventions: Biological: Autologous hematopoietic stem cell transplantation combined with CD19 CAR-T cells

INTERVENTIONS:
Biological: Autologous hematopoietic stem cell transplantation combined with CD19 CAR-T cells — The patient receives ECHOP chemotherapy or other chemotherapy regimens； G-CSF in the low cell stage mobilizes hematopoietic stem cells and freezes them for later use after collection； Autologous hematopoietic stem cells and prepared CD19 CAR-T cells are reinfused into the patient

SUMMARY:
Clinical Study on the Safety and Effectiveness of Autologous Hematopoietic Stem Cell Transplantation Combined With CAR-T Cells in the Treatment of Refractory and Relapsed Malignant Lymphoma

DETAILED DESCRIPTION:
Current studies have shown that under standard treatment, patients with large masses and high-grade DLBCL have a poor prognosis. Data from major centers around the world on CAR-T cell treatment of relapsed and refractory B-cell NHL show that CAR-T treatment of relapsed and refractory B-cell NHL has a low complete remission rate but a low recurrence rate after remission.Therefore, new treatment options are urgently needed to achieve long-term relief.

CD19 CAR-T therapy as a consolidation therapy after high-dose melphalan and autologous hematopoietic stem cell transplantation has been used in a refractory MM patient at the University of Pennsylvania, and good research progress has been made. Craig S et al. studied the safety and effectiveness of CD19 CAR-T cell therapy after high-dose chemotherapy and autologous stem cell transplantation HDT-ASCT. The object of the study was relapsed and refractory non-Hodgkin's lymphoma, with 2-year progression-free survival ( PFS) is 30%.

Therefore, autologous hematopoietic stem cell transplantation combined with CAR-T cell therapy is expected to improve the complete remission rate and long-term survival rate. In summary, the center intends to apply for a clinical trial of autologous hematopoietic stem cell transplantation combined with CAR-T cells for the treatment of refractory and relapsed non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female, 18-75 years old (including the threshold value); 2. According to the 2016 WHO classification criteria for lymphocytic tumors, histologically confirmed include: DLBCL (NOS); follicular lymphoma, chronic lymphocytic leukemia/small lymphocytic lymphoma transformed DLBCL, and PMBCL and high-grade B-cell lymphoma Subject.

  3.R/R B-NHL (conform one of the following conditions)
  1. The subject did not remission or relapsed after receiving second-line or higher-line chemotherapy
  2. Primary resistance
  3. The subject relapsed after receiving autologous hematopoietic stem cell transplantation

     Exclusion Criteria:
* Subjects with any of the following exclusion criteria were not eligible for this trial:

  1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
  2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
  3. Pregnant (or lactating) women;
  4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
  5. Active infection of hepatitis B virus or hepatitis C virus;
  6. Those who have used any gene therapy products before.
  7. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
  8. Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
  9. Those who suffer from other uncontrolled diseases are not suitable to join the study;
  10. HIV infection;
  11. Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate | Up to 30 months
  the number of response patients/the number of total patients
Incidence of treatment-emergent adverse events (TEAEs) | 24 months after cell infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Overall response rate(ORR) | Month 1,3,6,12,18and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 1,3,6,12,18and 24
Progression-free survival (PFS) | Month 6,12,18and 24
  Assessment of PFS at Month 6,12,18and 24
Overall survival (OS) | Month 6,12,18and 24
  Assessment of OS at Month 6,12,18and 24
Duration of response(DOR) | Month 6,12,18and 24
  Assessment of OS at Month 6,12,18and 24

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China